CLINICAL TRIAL: NCT02226796
Title: Effects of a Combination of Transcranial Direct Stimulation (tDCS) and Behavioral Intervention in Non-fluent Aphasia
Brief Title: Transcranial Direct Stimulation (tDCS) and Behavioral Intervention in Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1506M73043
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Aphasia
Keywords: Broca's Aphasia; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Aphasia; Aphasia, Broca | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Prime Condition (Active Comparator): The primed (PRIME) condition is an intervention that will consist of presentation of a-tDCS for 20 minutes to the dorsolateral prefrontal cortex prior to 40 minutes of behavioral naming treatment, while the subject sits comfortably in a chair.
  Interventions: Device: Transcranial direct current stimulation
- Non-Prime Condition/Control (Active Comparator): The non-primed (NON-PRIME) condition, or sham controlled, is an intervention that will consist of presentation of sham tDCS to the dorsolateral prefrontal cortex for 20 minutes prior to 40 minutes of behavioral naming treatment, while the subject sits comfortably in a chair.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation (tDCS) is a non-invasive neuromodulation tool that presents a low current that induces bi-directional polarity-dependent changes in the cortex to facilitate focal, prolonged shifts in cortical excitability at or around the time stimulation is provided. Anodal tDCS (a-tDCS), in which the positively charged electrode is placed over the targeted cortical region, has been shown to increase cortical excitability (upregulation), similar to long-term potentiation (LTP). Combining a-tDCS with behavioral-based approaches has been suggested to enhance the learning process and increase the likelihood of retention.

SUMMARY:
We hypothesize patients who have difficulty with word recall (naming pictures) due to a stroke will experience greater benefit in word recall after receiving a combination of transcranial direct current stimulation (tDCS) and traditional behavioral treatment. This study will investigate the effects of the timing of tDCS in relationship to the behavioral treatment to determine the most optimal protocol. Transcranial direct current stimulation involves placing two electrodes on your scalp and sending a very small electrical current to excite the brain cells of the target site.

DETAILED DESCRIPTION:
Specific Aims Aim 1: Identify and quantify the effects of a-tDCS to the left dorsolateral prefrontal cortex (DLPFC) in conjunction with intensive behavioral treatment on naming in non-fluent aphasia. a-tDCS (2mA for 20 minutes) will be applied over the left DLPFC with cathode over the right orbit. Pre and post treatment behavioral measures of naming and working memory will be used to quantify and compare differences. Hypothesis 1: a-tDCS will result in improvements in naming accuracy, naming response times, and working memory (WM) in participants with non-fluent aphasia.

Aim 2: Compare the effects of a-tDCS applied to the left DLPFC before behavioral treatment to during behavioral treatment in non-fluent aphasia. a-tDCS (2mA for 20 minutes) will be applied over the left DLPFC with cathode over the right orbit. Pre and post treatment behavioral measures of naming and working memory will be used to quantify and compare functional differences between conditions. Hypothesis 1: a-tDCS to the DLPFC during treatment will result in a greater improvement of naming accuracy, naming response time and WM in participants with non-fluent aphasia.

Significance The findings from the proposed study will lay the foundation for a larger clinical trial which will in turn have a significant impact on individuals with aphasia given that naming deficits are a common symptom in this population. As the presence of naming deficits has a negative relationship to emotional well-being and functional communication 26-30, treatment that improves naming deficits will positively influence quality of life in many of these individuals. The approach taken to remediate naming deficits in aphasia is to treat impaired WM systems on the premise that certain cognitive processes underlie linguistic functions in aphasia. This approach represents a departure from most behavioral-based naming treatment approach, but reflects a growing recognition that WM systems in individuals with aphasia impact their linguistic performance 5, 31. The addition of a-tDCS as a neuromodulation tool to increase cortical excitability (upregulate) the working memory center to target naming is a novel approach. In addition, this study will further elucidate the optimal timing of a-tDCS in order to achieve the most beneficial outcomes, which have not yet been reported. These findings, along with other related studies, will shape future clinical practice guidelines as more studies adopt a concurrent cognitive-linguistic approach to treat linguistic deficits in aphasia.

Design & Methodology Participants. Four individuals with aphasia will be recruited. These participants must meet the following inclusionary/exclusionary criteria: a) completion of high school or GED; b) normal or corrected-to-normal vision; c) adequate hearing acuity for 1:1 conversational exchanges; d) use of English as primary language; e) a vascular lesion in the dominant left hemisphere verified by an MRI scan within six months of the start of the study. These participants must also meet the following exclusionary criteria: a) no previous history of neurological- or psychiatric-based illnesses or disease, language or learning disabilities, or alcohol/substance abuse; b) no history of seizures; c) no metal implants in the head (except dental fillings); d) no lesion in the left DLPFC confirmed by MRI; e) no current pregnancy. Pre-Test Behavioral Measures. Participants will be seen between 2-3 sessions to undergo comprehensive cognitive-linguistic testing prior to initiation of treatment. Testing will take place at the University of Minnesota (UMN) Clinical Translational Science Institute (CTSI). Behavioral test measures will include the WAB 32 in order to obtain the WAB Aphasia Quotient (WAB AQ), Boston Naming Test (BNT) 33 and the Apraxia Battery for Adults (ABA-2) 34. The WAB AQ will provide a general classification of aphasia subtype, scores from the BNT will provide the level of severity of naming impairment, and ABA-2 performance will be used to assess severity of apraxia of speech (AoS). To assess the integrity of the phonological store, participants will be tested for the effects of phonological similarity using both auditory and visual presentation 35, 36. To assess the integrity of subvocal rehearsal processes, participants will be tested for the effects of word length on both auditory and visual span 37; the effects of articulatory suppression on recall performance 37, 38; and rhyme judgments 39-41. Protocols that have been adapted for individuals with aphasia will be followed42-45. These tests will be used to distinguish behavioral evidence of deficient subvocal rehearsal processes from deficient phonological short-term store. Individuals with a range of moderate to moderately severe nonfluent aphasia, a range of moderate to moderately severe anomia, and a range of mild to no AoS will be chosen for the study. Baseline probes will also be obtained prior to the initiation of the study. Stability of baseline performance, defined as no more than 20% difference between scores,will be obtained over three consecutive sessions in order to establish experimental control. Post-Test Behavioral Measures. Participants will also be seen for post-treatment testing following the implementation of the treatment protocol. Testing will take place in the participant's home. Post-treatment behavioral measures will include BNT, the ABA-2, WM tasks, and naming treatment and control items. It is anticipated that only one session will be needed for post-treatment testing. An adverse events survey will also be provided to assess the participant's level of discomfort during use of tDCS. tDCS Protocol. Each participant will be seated comfortably in a chair. A swim cap will be placed on the participant's head to identify cranial landmarks for accurate electrode placement. The area referred to as F3 by the International 10/20 system for electroencephalogram electrode placement46 has been established as the optimal location for targeting the left DLPFC25, 47-49. The F3 region will be located by marking the vertex (the midpoint between left and right tragus and midpoint between nasion and inion), measuring the head circumference. When these measurements are entered into the Beam F3 Locator Software50, additional values are provided to reliably identify the location of F3. Once F3 has been established, two saline soaked surface sponge electrodes (352cm) will be prepared and placed. For optimal anodal stimulation to the DLPFC, the anode will be placed over F3 and the cathode will be placed over the right supraorbital region23, 24, 47, 48. A current of 2mA will be delivered for 20 minutes 24 by a multichannel transcranial current stimulator (Starstim, Neuroelectrics Corporation; Cambridge, MA). a-tDCS will be applied before and during behavioral treatment in the design specified below.

Treatment Design. Two treatment conditions will be presented in a counter-balanced order in a cross-over design. The non-prime (NONPRIME) condition will consist of 40 minutes of naming treatment only, followed by an additional 20 minutes of concurrent naming treatment with a-tDCS. The primed (PRIME) condition will consist of presentation of a-tDCS for 20 minutes prior to naming treatment, while the subject sits quietly and comfortably in a chair. After the 20-minute priming period, the a-tDCS will be removed and the participant will receive naming treatment for 60 minutes. Both conditions will be presented over four consecutive days. Two participants will receive NON-PRIME-PRIME sequence, with a one-month washout period between the two conditions. Two other participants will receive PRIME-NON-PRIME sequence, with a one-month washout period between the two conditions. Naming reaction time will be immediately evaluated after each treatment day.

ELIGIBILITY:
Inclusion Criteria:

* completion of high school or GED, normal or corrected-to-normal vision, adequate hearing acuity for 1:1 conversational exchanges, use of English as primary language, a vascular lesion in the dominant left hemisphere verified by an MRI scan within six months of the start of the study

Exclusion Criteria:

* no previous history of neurological- or psychiatric-based illnesses or disease, language or learning disabilities, or alcohol/substance abuse; no history of seizures; no metal implants in the head (except dental fillings); no lesion in the left DLPFC confirmed by MRI; no current pregnancy.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharyl A Samargia, PhD, Principal Investigator — University of Minnesota and University of Wisconsin
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
The protocol for sharing individual participant data with other researchers has not yet been determined as data collection is in progress.

RESULTS

PARTICIPANT FLOW:
Groups:
- Primed tDCS Condition First, Then Non-Prime Condition: The primed (PRIME) condition is an intervention that will consist of presentation of a-tDCS for 20 minutes to dorsolateral prefrontal cortex prior to 40 minutes of behavioral naming treatment, while the subject sits comfortably in a chair.
  The non-primed (NONPRIMED) condition, or sham/control is an intervention that will consist of presentation of sham tDCS for 20 minutes to dorsolateral prefrontal cortex prior to 40 minutes of behavioral naming treatment, while the subject sits comfortably in a chair.
- Non-Prime Condition First, Then Primed Condition: The non-primed (NONPRIMED) condition, or sham/control is an intervention that will consist of presentation of sham tDCS for 20 minutes to dorsolateral prefrontal cortex prior to 40 minutes of behavioral naming treatment, while the subject sits comfortably in a chair.
  The primed (PRIME) condition is an intervention that will consist of presentation of a-tDCS for 20 minutes to dorsolateral prefrontal cortex prior to 40 minutes of behavioral naming treatment, while the subject sits comfortably in a chair.
Period: First Intervention Phase (Week 1)
Arm/Group | Primed tDCS Condition First, Then Non-Prime Condition | Non-Prime Condition First, Then Primed Condition
Started | 2 | 1
Baseline Assessment | 2 | 1
Follow Up Assessment | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0
Period: Washout (Weeks 2-5)
Arm/Group | Primed tDCS Condition First, Then Non-Prime Condition | Non-Prime Condition First, Then Primed Condition
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0
Period: Second Intervention Phase (Week 6)
Arm/Group | Primed tDCS Condition First, Then Non-Prime Condition | Non-Prime Condition First, Then Primed Condition
Started | 2 | 1
Baseline Assessment | 2 | 1
Follow Up Assessment | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham Controlled tDCS Combined With Behavioral Naming Treatment: The primed (PRIME) condition is an intervention that will consist of presentation of a-tDCS for 20 minutes prior to 40 minutes of behavioral naming treatment, while the subject sits comfortably in a chair.
  The non-prime (NONPRIME) condition, sham/control is an intervention that will consist of 40 minutes of naming treatment only, followed by an additional 20 minutes of concurrent naming treatment with a-tDCS.
  Behavioral measures taken include: working memory, naming reaction time and naming accuracy
Arm/Group | Sham Controlled tDCS Combined With Behavioral Naming Treatment
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.33 (18.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3
Working Memory [Mean (Standard Deviation); unit: units on a scale] — During the Working Memory battery, participants completed 12 auditory only or auditory & visual computer-based recall tasks. Twelve subset scores were calculated. Total score is calculated as sum of subtest scores and ranges from 0-520 with higher scores indicating greater working memory.
  The following auditory and auditory/visual subtests have a possible scoring range between 0-40: phonologically similar and dissimilar word span, word length (short and long) and word span The digit span (auditory and visual/auitory) has scoring range of 0-60. Higher values represent better performance.
  units on a scale
    AudioVisual_LongWordLength | 16.33 (12.97)
    AudioVisual_ShortWordLength | 17 (12.72)
    AudioVisual_WordSpan | 18.66 (11.58)
    Visual_DigitSpan | 8.66 (3.39)
    Visual_PhonologicallySimilarWords | 7.66 (6.12)
    Visual_PhonologicallyDissimilarWords | 12.5 (3.5)
    Visual_LongWordLength | 6 (4.24)
    Visual_ShortWordLength | 9.66 (5.79)
    Visual_WordSpan | 11 (3.26)
    Total Score | 148 (102.30)
Western Aphasia Battery Score [Mean (Standard Deviation); unit: units on a scale] | 52.23 (12.30)
Boston Naming Test [Mean (Standard Deviation); unit: units on a scale] | 12 (0.81)
Naming Reaction Time [Mean (Standard Deviation); unit: time in milliseconds] — Participants are shown one or 3 possible banks of pictures balanced for phonemic complexity which are randomly assigned to prevent learning effect. Each bank contains 10* items. Time to recall is measured using a stop watch. The mean time to recall across all items is calculated and reported in milliseconds. The smaller the number, the faster / better the reaction time is.
  time in milliseconds | 2986.03 (1260.48)
Naming Accuracy [Mean (Standard Deviation); unit: units on a scale] — Participants are shown one or 3 possible banks of pictures balanced for phonemic complexity which are randomly assigned to prevent learning effect. Each bank contains 10* items. Each trial is scored by an examiner as accurate (1) or inaccurate (0). The sum* of all trials is calculated. Total scores range from 0-10* with higher scores indicating better naming accuracy/performance.
  units on a scale | 4.48 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Naming Reaction Time
Description: Participants are shown one or 3 possible banks of pictures balanced for phonemic complexity which are randomly assigned to prevent learning effect. Each bank contains 15 items. Time to recall is measured using a stop watch. The mean time to recall across all items is calculated and reported in milliseconds. The smaller the number, the faster / better the reaction time is.
Time Frame: 40 minutes
Population: This is a single subject cross over design where all three participants received both prime and non-prime condition
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Prime Condition | Non-Prime Condition/Control
Number analyzed (Participants) | 3 | 3
milliseconds | 1829.11 (643.40) | 3345.97 (1428.38)

2. Primary Outcome: Naming Accuracy
Description: Participants are shown one of 3 possible banks of pictures balanced for phonemic complexity which are randomly assigned to prevent learning effect. Each bank contains 15 items. Each trial is scored by an examiner as accurate (1) or inaccurate (0) based on articulatory accuracy of the participant's response. The average of all trials is calculated for each participant. Total scores range from 0-15 with higher scores indicating better naming accuracy/performance.
Time Frame: 40 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prime Condition | Non-Prime Condition/Control
Number analyzed (Participants) | 3 | 3
units on a scale | 5.95 (2.59) | 6.044 (2.32)

3. Secondary Outcome: Boston Naming Test
Description: The Boston Naming Test contains 60 line drawings of objects ranging from very common objects to less familiar. The examiner scores each item + or - according to scoring procedures. Total scores are calculated by adding up the number correct. Scores range from 0 to 60. Higher scores indicate greater ability to name objects.
Time Frame: 30 minutes
Population: The Co-PI collected data using the Boston Naming Test at baseline (before either prime or non-prime condition) and after both conditions were complete. No BNT data was collected between the two conditions, therefore we cannot determine the impact of the prime condition on BNT scores. Flawed execution of this outcome measure.
Arm/Group | Prime Condition | Non-Prime Condition/Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Western Aphasia Battery Total Score
Description: The Western Aphasia Battery, a standardized assessment of language for individuals with aphasia, contains 32 short tasks. Each task has a separate scoring scheme yielding 8 sub-scores. Total score range from 0-100 with lower scores indicating greater aphasia severity. A score between 0-25 is very severe aphasia, 26-50 is severe aphasia, 51-75 is moderate aphasia, and 76-above is mild aphasia.
Time Frame: 60 minutes
Population: The Co-PI collected data using the Western Aphasia Battery at baseline (before either prime or non-prime condition) and after both conditions were complete. No BNT data was collected between the two conditions, therefore we cannot determine the impact of the prime condition on WAB scores. Flawed execution of this outcome measure.
Arm/Group | Prime Condition | Non-Prime Condition/Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Working Memory Total Score
Description: During the Working Memory battery, participants complete 12 auditory only or auditory & visual computer-based recall tasks. Twelve subset scores are calculated. Ten subtest ranges from 0-40 and 2 range from 0-60. Total score is calculated as sum of subtest scores and ranges from 0-520 with higher scores indicating greater working memory.
Time Frame: 2 months
Population: The Co-PI collected data using the working memory assessment at baseline (before either prime or non-prime condition) and after both conditions were complete. No BNT data was collected between the two conditions, therefore we cannot determine the impact of the prime condition on working memory scores. Flawed execution of this outcome measure.
Arm/Group | Prime Condition | Non-Prime Condition/Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 months
Description: Each participant was asked if they experienced headache or itchy/tingly sensation at site of stimulation during and/or after tDCS sessions.
Groups:
- Primed tDCS Condition: The primed (PRIME) condition is an intervention that will consist of presentation of a-tDCS for 20 minutes to dorsolateral prefrontal cortex prior to 40 minutes of behavioral naming treatment, while the subject sits comfortably in a chair. Naming reaction time and accuracy will be measured as well as working memory.
- Non-Prime Condition: The non-primed (NONPRIMED) condition, or sham/control is an intervention that will consist of presentation of sham tDCS for 20 minutes to dorsolateral prefrontal cortex prior to 40 minutes of behavioral naming treatment, while the subject sits comfortably in a chair. Naming reaction time and accuracy will be measured as well as working memory.
Arm/Group | Primed tDCS Condition | Non-Prime Condition
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT02226796/Prot_SAP_000.pdf